CLINICAL TRIAL: NCT02773589
Title: Prospective Evaluation of a New Approach to Perform an Esophageal Myotomy: the Transesophageal Submucosa Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5368
Record Dates: First submitted 2016-05-09; First posted 2016-05-16 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2016-05

CONDITIONS: Esophagus Achalasia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peroral endoscopic myotomy (Experimental)
  Interventions: Procedure: Peroral endoscopic myotomy

INTERVENTIONS:
Procedure: Peroral endoscopic myotomy — Peroral endoscopic myotomy

SUMMARY:
Achalasia is an esophagus motor disability characterized by a lack of relaxation of the lower esophageal sphincter (LES) to deglutition. Myotomy is the gold standard surgical technique allowing to cure this pathology. In this study, investigators are using a new endoluminal technique of myotomy, innovative and less invasive, called POEM (PerOral Endoscopic Myotomy). This technique does not require any cutaneous incision.

Mini-invasive surgery is more and more associated to endoscopy. The practice was initiated by the accession of natural orifice transluminal endoscopic surgery (NOTES). In this context, the introduction of the POEM technique seems to be an original approach and a natural evolution to a new generation of surgical endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Esophagus achalasia
* Confirmed by esophageal manometry
* Requiring surgical care
* No contraindication to general anesthesia
* BMI under 40 kg/m²
* Ability to give an informed consent
* Candidate to elective Heller's myotomy
* Affiliation to a social security system
* Signed and informed consent

Exclusion Criteria:

* Advanced esophageal dilatation (sigmoid megaesophagus)
* Previous mediastinal or esophageal surgery
* Contraindication to esophagogastroduodenoscopy (EGD)
* Contraindication to general anesthesia
* BMI above 40 kg/m²
* Infectious esophagitis (e.g. candidiasis)
* Psychiatric context unsuitable with an experimental protocol
* Allergy to beta-lactam
* Contraindication to endoscopy (esophageal stenosis, suspicion of digestive perforation, state of shock, severe anemia, cardiorespiratory failure or severe metabolic disorders)
* Contraindication to monitored pneumoperitoneum (cardiorespiratory failure or severe metabolic disorders)
* Inability to give an informed consent (emergency situations, misunderstanding…)
* Patient in custody
* Patient under guardianship
* Pregnancy or breastfeeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The safety assessment will be based on the reading of all surgical intraoperative complications | 6 months post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Silvana PERRETTA, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- University Hospital, Strasbourg, france, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No